CLINICAL TRIAL: NCT02169830
Title: A Prospective Randomized Cross-over Trial of Nortryptyline and Topiramate in the Initial Treatment of Vestibular Migraine.
Brief Title: Trial of Nortriptyline and Topiramate in the Initial Treatment of Vestibular Migraine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Anthony A. Mikulec, MD, Associate Professor, St. Louis University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24482_ Vest_Migraine
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Migraine Disorders
Keywords: vestibular migraines, nortriptyline and topiramate
MeSH Terms: conditions — Migraine Disorders | interventions — Nortriptyline; Topiramate; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- nortriptyline (Active Comparator): If after four (4) weeks of diet modification, patients are still experiencing migraines, they may be randomized to nortriptyline for eight (8) weeks. If still experiencing symptoms, they will receive topiramate for eight (8) weeks.
  Interventions: Drug: nortriptyline
- topiramate (Active Comparator): If after four (4) weeks of diet modification, patients are still experiencing migraines, they may be randomized to topiramate for eight (8) weeks. If still experiencing symptoms, they will receive nortriptyline for eight (8) weeks.
  Interventions: Drug: Topiramate
- diet modification (Other): Participants will begin with diet modification for four (4) weeks.
  Interventions: Behavioral: Diet Modification

INTERVENTIONS:
Drug: nortriptyline — The nortriptyline will be given in an escalating fashion, starting at 25 mg PO qhs for 2 weeks, followed by 50 mg PO qhs for 2 weeks, and finally 75 mg PO qhs. Patients will be encouraged to use the lowest effective dose and to self-titrate their medication.
  Other Names: Nortriptyline HCI
  Arms: nortriptyline
Drug: Topiramate — Topiramate dosing will be 25 mg PO qhs for 1 week, followed by 25 mg BID for 1 week, followed by 25 mg in the morning and 50 mg qhs for 1 week, and finally 50 mg BID
  Other Names: Topamax
  Arms: topiramate
Behavioral: Diet Modification — Emphasis will be given to cessation of known migraine triggers such as caffeine, sodas, chocolates, alcohol (especially red wine) and aged cheeses. Patients who have complete control of their symptoms with diet and behavior modification alone will be followed for a total of 4 months to determine the durability of symptom relief.
  Arms: diet modification

SUMMARY:
The investigators' study plans to randomize treatment naive patients with vestibular migraine to an 8 week trial of an escalating dose of either nortriptyline or topiramate followed by an 8 week crossover to the other drug if patient is willing, if patient wants to stay on first medication we will just continue to follow. During the first 8 weeks if there is an intolerance to the first drug they can be switched to the other drug at any point and then followed on that medication for the remainder of the study. Response to therapy will be quantified by the Migraine Specific Quality of Life (MSQ) and Dizziness Handicap Inventory (DHI) administered at multiple time points during the study. Three groups of patients that will be eligible for the study will include 1)Patients with Neuhauser dVM; 2)Patients with pVM; and 3) Patients with dizziness that falls outside the Neuhauser criteria (non-Neuhauser vestibular migraine or nNVM).

The investigators' hypothesis is that even patients with dizziness outside of the Neuhauser dVM and pVM spectrum will respond to treatment for vestibular migraine, and thus likely have migraine as a cause of their dizziness. Previous research by our group has suggested that such patients do in fact respond to migraine therapy1. A second goal of the study is to evaluate the comparative efficacy of nortriptyline and topiramate in the treatment of these three subgroups of patients with vestibular migraine.

DETAILED DESCRIPTION:
After identification and trial entry, we will complete intake questionnaire to determine what type of vestibular migraine category the patients qualify for, a standard of care office visit with history and physical (Standard of Care) to review symptoms and previous treatment, patients height and weight (standard of care) will be obtained. Patients will complete a standard of care audiology assessment, and the following questionnaires: MSQ (Migraine Symptom Questionnaire) Version 2.1, DHI (Dizziness Questionnaire) , C-SSRS (Columbia Suicide Severity Rating Scale) and the MoSQ (Motion Sensitivity Questionnaire). All drug naive patients will undergo a one month lead in of treatment involving dietary and behavioral control of migraine. Emphasis will be given to cessation of known migraine triggers such as caffeine, sodas, chocolates, alcohol (especially red wine) and aged cheeses. Patients who have complete control of their symptoms with diet and behavior modification alone will be followed for a total of 4 months to determine the durability of symptom relief. Patients who fail behavior modification during the 2 to 4 month time point can chose to enter the drug treatment portion of the study, as defined below.

At the one month point, patients will be brought into the clinic for a office visit with history, physical, and weight checked and will complete MSQ V2.1, DHI, C-SSRS and the MoSQ, then will be randomization to either nortriptyline or topiramate will occur. Randomization will occur by opening the lowest numbered of a stack of envelopes which will contain a randomly preselected card indicating which drug is to be used. The nortriptyline will be given in an escalating fashion, starting at 25 mg PO qhs for 2 weeks, followed by 50 mg PO qhs for 2 weeks, and finally 75 mg PO qhs. Patients will be encouraged to use the lowest effective dose and to self-titrate their medication. Topiramate dosing will be 25 mg PO qhs for 1 week, followed by 25 mg BID for 1 week, followed by 25 mg in the morning and 50 mg qhs for 1 week, and finally 50 mg BID. Patients will be allowed considerable leeway in adjusting their dosage and will be encouraged to stay on the lowest effective dose. Medication will be provided open label to the patient and paid for through the patients' insurance, as this intervention falls within current standard practice, and is not investigational.

After two, three and four months on drug patients will be brought into the clinic for a office visit with history, physical, and weight checked and will complete MSQ V2.1, DHI, C-SSRS and the MoSQ, then patients will be offered the opportunity to switch to the other drug. Those patients who wish to switch drugs will first be weaned off their current drug over a one week time period. Patients who elect to stay on their initial drug will be followed for a total of four months. Patients who opt for trial of a second drug will then be started on the second drug via a self-titrating protocol as described above and followed on that drug for up to 4 months.

The investigators' clinical experience has shown that on occasion patients will refuse to take more than a few doses of nortriptyline or topiramate due to intolerable side effects. Such patients will be allowed to immediately initiate therapy with the other drug. The medication change can be done with a phone call to their pharmacy without an office visit, as is done in standard of care. Also, patients who already follow a rigorous migraine diet will be allowed to enter the drug treatment phase immediately. In our experience, such patient make up less than 5% of the population that presents for treatment of vestibular migraine.

The response to therapy will be assessed during monthly visits with the use of the MSQ, DHI and MoSQ questionnaires. Patients will be provided compensation for participating in the study. $60 dollars will be paid to each patient for each month that they participate in the study. Our goal is to recruit 100 patients over the span of one year.

Data which will be collected include age, sex, height, weight, body mass index (BMI), prior head MRI or CT, results of vestibular testing, family history of migraine. A careful history will focus on vestibular migraine comorbidities such as visual scotoma, ability to ride in the back seat of a car, and history of "sinus pain".

Patients will be identified as having one of three subtypes of vestibular migraine, based on their symptoms and history as obtained during their initial visit.

Criteria for Neuhauser definite vestibular migraine (dVM): (Neuhauser, 2009):

1. Episodic vestibular symptoms of at least moderate severity.
2. Current of previous history of migraine according to the 2004 criteria of the International Headache Society (IHS)
3. One of the following migrainous symptoms during 2 or more attacks of vertigo: migrainous headache, photophobia, phonophobia, visual aura, or other aura
4. Other causes ruled out by appropriate investigations

Criteria for probable vestibular migraine (pVM):

1. Episodic vestibular symptoms of at least moderate severity
2. One of the following A. current or previous history of migraine according to the 2004 criteria of the IHS B. migrainous symptoms during vestibular symptoms C. migraine precipitants of vertigo in > 50% of attacks: food triggers, sleep irregularities, or hormonal change D. Response to migraine medications in more than 50% of attacks
3. Other causes ruled out by appropriate investigations

Criteria for (non-Neuhauser vestibular migraine or nNVM) will include those patients who do not fit the criteria for dVM and pVM but are felt by the investigator to have underlying migraine as a possible cause of their dizziness. This includes patients with a remote history of migraines, those with visual auras without headache, those with recurring self-described "sinus pain" and those with significant motion intolerance, either to their own head motion or motion in their surroundings.

Due to know drug interactions, patients taking the following medications will be excluded.

Nortriptyline: monoamine oxidase inhibitors (MAO) such as phenelzine. Patients on oral contraceptives will be asked to use a secondary method as nortriptyline can reduce the effectiveness of oral contraceptives.

Topiramate: acetazolamide (kidney stones), digoxin

An electronic health record (EPIC) will be used for secure collection of all patient data. Questionnaires filled out by patients will be scanned into EPIC.

A sample size of 100, which nets 90 subjects into the randomized medication trial (two equal groups of 45 subjects each), yields a power of 82% to detect a difference in patient-reported effectiveness/acceptability between the nortriptyline and topiramate groups after two months of medication use. This sample size estimate assumes 60% of subjects using nortriptyline report it as effective/acceptable, in contrast to half as many subjects (or 30%) using topiramate. The power calculation is based on a two-sized Z-test with pooled variance and targeted significance level (alpha) of 0.05. The expected difference in outcome between the two groups is based on our prior research (Mikulec, 2012).

Adverse effects of the two drugs will be assessed. Specifically, the following known side effects will be asked about and recorded.

Nortriptyline: somnolence, weight gain, dry mouth, blurred vision Topiramate: Weight loss, parasthesias, forgetfulness, nausea, diarrhea, fatigue

The subjects will be allowed to maintain therapy or taper off the drugs. It is anticipated that those that derive benefit from the drugs will choose to stay on them. All patients will have the option of remaining under our care outside of the study.

ELIGIBILITY:
Inclusion Criteria:

-Men and women aged 18 to 70 with untreated vestibular migraine variant as diagnosed by history.

Exclusion Criteria:

* Patients with allergies to nortriptyline or topiramate and their analogs or medication interactions that preclude their use.
* Patients under the care of a psychiatrist.
* Patients who are pregnant or trying to become pregnant.
* Patients taking more than 5 prescription medications.
* Patients with cancer.
* Patient has a history of immunodeficiency.
* Patient has a history of substance abuse within the preceding 6 months prior to screening.
* Patient has used an investigational drug or device in the the 3 months prior to screening.
* Patient is using marijuana for medical or other uses.
* Patient has any other clinically significant illness or medical condition that, in the investigator's opinion, would prohibit the subject from participating in the study.
* Patient with traumatic brain injury.
* Patients taking Nortriptyline, MAOIs
* Patients with liver or kidney dysfunction or glaucoma

Due to know drug interactions, patients taking the following medications will be excluded.

Nortriptyline: monoamine oxidase inhibitors (MAO) such as phenelzine. Patients on oral contraceptives will be asked to use a secondary method as nortriptyline can reduce the effectiveness of oral contraceptives.

Topiramate: acetazolamide (kidney stones), digoxin

Exclude subjects with liver dysfunction, kidney dysfunction and glaucoma (per the risks associated with topiramate).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-08-22 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A Mikulec, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 patients were screened between August 2014 and November 2016.
Pre-assignment Details: 33 of 35 began the study with diet modification. 2 subjects who were fully consented dropped out of the study before randomization.
Groups:
- Nortriptyline: Diet modification - nortriptyline and then if necessary topiramate
  nortriptyline: The nortriptyline will be given in an escalating fashion, starting at 25 mg PO qhs for 2 weeks, followed by 50 mg PO qhs for 2 weeks, and finally 75 mg PO qhs. Patients will be encouraged to use the lowest effective dose and to self-titrate their medication.
- Topiramate: Diet Modification topiramate and then nortriptyline if necessary
  Topiramate: Topiramate dosing will be 25 mg PO qhs for 1 week, followed by 25 mg BID for 1 week, followed by 25 mg in the morning and 50 mg qhs for 1 week, and finally 50 mg BID
Period: Diet Intervention (4 Weeks)
Arm/Group | Nortriptyline | Topiramate | Diet Modification
Started | 0 | 0 | 33
Completed | 0 | 0 | 32
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Second Intervention (8 Weeks)
Arm/Group | Nortriptyline | Topiramate | Diet Modification
Started | 12 | 5 | 0
Completed | 9 | 0 | 0
Not Completed | 3 | 5 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 5 | 0
Period: Third Intervention (8 Weeks)
Arm/Group | Nortriptyline | Topiramate | Diet Modification
Started | 0 | 4 (These four subjects were randomized to Diet first Topiramate second, and Nortriptyline third. No subjects from this group were weaned and moved to Nortriptyline.) | 0
Completed | 0 | 2 | 0
Not Completed | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects started study with diet modification. Of the 35 consented subjects the completion breakdown is as follows:
  18 subjects diet modification only; 6 subjects diet modification then nortriptyline; 9 subjects diet modification then topiramate; 2 subjects consented and were no show for all other study visits.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nortriptyline | Topiramate | Diet Modification | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical — Data was not intended to be nor was it collected. Population: Data was not intended to be nor was it collected.
Age, Continuous [unit: years] — Data was not intended to be nor was it collected. Population: Data was not intended to be nor was it collected.
Sex: Female, Male — Data was not intended to be nor was it collected. Population: Data was not intended to be nor was it collected.
Race (NIH/OMB) — Data was not intended to be nor was it collected. Population: Data was not intended to be nor was it collected.
Region of Enrollment [unit: participants] — Data was not intended to be nor was it collected. Population: Data was not intended to be nor was it collected.

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Comparative Effectiveness of Migraine Diet, Nortriptyline and Topiramate
Description: Changes in Migraine Specific Quality of LIfe (MSQ) and Dizziness Handicap Inventory (DHI) between groups
Time Frame: one year
Population: No data was collected.
Arm/Group | Nortriptyline | Topiramate | Diet Modification
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored until subjects dropped, were lost to follow up, or completed the study, an average of 1 quarterly per participant.
Arm/Group | Nortriptyline | Topiramate | Diet Modification
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/33
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT02169830/Prot_SAP_000.pdf